CLINICAL TRIAL: NCT05779917
Title: Mesothelin/GPC3/GUCY2C Targeted CAR-T for Immunotherapy of Pancreatic Cancer: Phase I Clinical Trial
Brief Title: Mesothelin/GPC3/GUCY2C-CAR-T Cells Against Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital of Guangzhou Medical University (Other)
Collaborators: Fapon Biotherapy Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZZFC004CAR-018
Record Dates: First submitted 2023-03-10; First posted 2023-03-22 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Pancreas Cancer; CAR-T Cell Therapy; Mesothelin; Solid Tumor, Adult
Keywords: Pancreas Cancer; CAR-T; Mesothelin; Solid Tumor
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Immunotherapy, Adoptive

STUDY DESIGN:
Intervention Model Description: Use engineered CAR-T cells to kill cancer cells with mesothelin overexpression.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: CAR-T cells — Transfer CAR-T cells into patients for anti-ancer therapy.

SUMMARY:
The second generation of mesothelin targeted CAR-T cells that secret a fusion protein of IL21 and scfv against PD1 have been constructed and their anti-cancer function has been verified by multiple in vitro and in vivo studies. Clinical studies will be performed to test anti-cancer function of the CAR-T cells for immunotherapy of human cancer patients with Mesothelin expressions. In this phase I study, the safety, tolerance, and preliminary efficacy of the Mesothelin-CAR-T cell immunotherapy on human cancers will firstly be evaluated.

DETAILED DESCRIPTION:
1. Choose appropriate patients with advanced pancreatic cancer or other cancers, with written consent for this study;
2. Perform biopsy to determine the expression of Mesothelin of the tumors by western blotting or IHC;
3. Collect blood from the patients and isolate mononuclear cells, activate the T cells and transfect the T cells with Mesothelin targeting CAR, amplify the transfected T cells as needed, test the quality and killing activity of the CAR-T cells and then transfer them back the patients via systemic or local injections, and follow up closely to collect related results as required;
4. To enhance the killing capability, cotreatment the patients with PD1/PDL1/CTLA4 antibodies may be applied;
5. Evaluate the clinical results as needed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with advanced cancer that expresses Mesothelin protein; 2. Life expectancy >12 weeks; 3. Adequate heart, lung, liver, kidney, and blood function; 4. Available autologous transduced T cells with greater than or equal to 20% expression of Mesothelin-CAR determined by flow-cytometry and killing of Mesothelin-positive targets greater than or equal to 20% in cytotoxicity assay; 5. Informed consent explained to, understood by and signed by patient/guardian. Patient/guardian given copy of informed consent.

-

Exclusion Criteria:

1. Had accepted gene therapy before;
2. Severe virus infection such as HBV, HCV, HIV, et al;
3. Known HIV positivity;
4. Active infectious disease related to bacteria, virus,fungi,et al;
5. Other severe diseases that the investigators consider not appropriate;
6. Pregnant or lactating women;
7. Systemic steroid treatment (greater than or equal to 0.5 mg prednisone equivalent/kg/day);
8. Other conditions that the investigators consider not appropriate. -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-03-10 (Actual); Primary Completion 2029-03-10 (Estimated); Study Completion 2036-03-10 (Estimated)

PRIMARY OUTCOMES:
Number of Patients with Dose Limiting Toxicity | six months
  A dose limiting toxicity is defined as any toxicity that is considered to be primarily related to the Mesothelin-CAR T cells, which is irreversible, or life threatening or hematologic or non-hematologic Grade 3-5.

SECONDARY OUTCOMES:
Percent of Patients with best response as either complete remission or partial remission. | six months
  Response rates will be estimated as the percent of patients whose best response is either complete remission or partial remission by combining the data from the patients. To compare with historical data, a 95% confidence interval will be calculated for the response rate.
Median CAR-T cell persistence | Six years
  Median CAR-T cell persistence will be measured by quantitative rt-PCR.

CONTACTS AND LOCATIONS:
Overall Officials: Zhenfeng Zhang, MD, PhD, Principal Investigator — Second Affiliated Hospital of Guangzhou Medical University
Locations (1):
- The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No